CLINICAL TRIAL: NCT02073331
Title: A Post Market Observational Study to Obtain Additional Information on the Use of CorMatrix ECM for Pericardial Reconstruction
Brief Title: Obtain Additional Information on Use of CorMatrix ECM (Extracellular Matrix)
Acronym: RECON
Status: Completed | Type: Observational
Sponsor: Elutia Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-PR-1095
Record Dates: First submitted 2014-02-24; First posted 2014-02-27 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Coronary Disease
Keywords: Open heart surgery, cardiac repair
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CorMatrix ECM: Data collection for information on the use of CorMatrix ECM for pericardial reconstruction

SUMMARY:
The objective of the study is to actively gather additional information on the use of CorMatrix ECM for pericardial reconstruction.

DETAILED DESCRIPTION:
Up to 100 clinical sites will enroll subjects who have received CorMatrix ECM for pericardial reconstruction.

The following clinical data will be collected at a single post-operative visit:

* Demographic information
* Pre-operative risk factors
* Surgical procedure
* Blood transfusion information, if applicable
* Chest tube placement information
* Surgical complications
* Use of anticoagulation medication
* Cardiac related procedures since surgical procedure
* Device related adverse events

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have received CorMatrix ECM for pericardial reconstruction
* Sign an Informed Consent

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have received CorMatrix ECM for pericardial reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 1420 (Actual)
Dates: Start 2014-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Green, Study Director — Elutia Inc.
Locations (42):
- United States (42):
  - Cario-Thoracic Surgeons, P.C., Birmingham, Alabama
  - Cardiovascular Consultants, LTD, Glendale, Arizona
  - Phoenix Cardiac Surgery, Phoenix, Arizona
  - Southwest Heart & Lung, Phoenix, Arizona
  - University of Arizona Medical Center, Tucson, Arizona
  - Mercy Clinic Cardiac Thoracic & Vascular Surgery, Fort Smith, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Baptist Medical Center, Little Rock, Arkansas
  - Heart & Lung Surgical Specialties, Rancho Mirage, California
  - Stockton Cardiothoracic Surgical Medical Group, Stockton, California
  - Hartford Healthcare Medical Group, Hartford, Connecticut
  - Tenet Florida Physician Services, Delray Beach, Florida
  - South Florida Heart & Lung Institute, Doral, Florida
  - Cardiothoracic & Vascular Surgical Associates, Jacksonville, Florida
  - David L. Galbut, MD & Associates, Miami, Florida
  - Palm Beach Gardens Medical Center, Palm Beach Gardens, Florida
  - Coastal Cardiovascular Surgeons, Panama City, Florida
  - Southern Cardiac & Vascular Associates, Tallahassee, Florida
  - Cardio Thoracic Vascular Surgery, Macon, Georgia
  - Community Health Network, Indianapolis, Indiana
  - Reid Hospital, Richmond, Indiana
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Health Systems, Detroit, Michigan
  - Western Michigan University Homer Stryker Medical Center School of Medicine for Clinical Research, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Magnolia Regional, Corinth, Mississippi
  - Baptist Cardiovascular Surgery, Jackson, Mississippi
  - St. Peter's Health Partners, Albany, New York
  - Triad Cardiac & Thoracic Surgeons, Greensboro, North Carolina
  - Wake Medical, Raleigh, North Carolina
  - Coastal Thoracic Surgical Associates, Wilmington, North Carolina
  - Novant Health Cardiothoracic Surgeons, Winston-Salem, North Carolina
  - TriStar Cardiovascular Surgery, Nashville, Tennessee
  - Advanced Cardiovascular & Thoracic Surgery, Nashville, Tennessee
  - Cardiothoracic & Vascular Surgeons, PA, Austin, Texas
  - Cardiothoracic Associates, Corpus Christi, Texas
  - Tung H. Cai, MD, PA, Denton, Texas
  - KPS Cardiovascular Surgery, Shenandoah, Texas
  - Mountain Star Cardiovascular Services, LLC, Salt Lake City, Utah
  - Carilion Cardiothoracic Surgery, Roanoke, Virginia
  - Thoracic & Cardiovascular Associates, Inc., Charleston, West Virginia

REFERENCES:
- [Derived] Rego A, Cheung PC, Harris WJ, Brady KM, Newman J, Still R. Pericardial closure with extracellular matrix scaffold following cardiac surgery associated with a reduction of postoperative complications and 30-day hospital readmissions. J Cardiothorac Surg. 2019 Mar 15;14(1):61. doi: 10.1186/s13019-019-0871-5. PMID 30876459

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CorMatrix ECM
Started | 1420
Completed | 1420
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CorMatrix ECM
Number analyzed (Participants) | 1,420
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 845
  >=65 years | 575
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 376
  Male | 1,044
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 118
  Not Hispanic or Latino | 1,302
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 158
  White | 1,088
  More than one race | 141
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 1,420
Pre-Operative Risk Factors [Number; unit: Risk factors]
  Hypertension | 1,138
  Hypercholesterolemia | 727
  Diabetes Mellitus | 531
  Smoking | 357
  Prior Myocardial Infarction | 242
  Congestive Heart Failure | 226
  Chronic Obstructive Pulmonary Disease | 158
  Prior Percutaneous Coronary Intervention | 126
  Chronic Renal Failure | 70
  Prior Cerebrovascular Accident | 60
Index Procedure [Count of Participants; unit: Participants]
  Isolated CABG | 923
  Valve Repair/Replacement | 300
  CABG & Valve Repair/Replacement | 136
  Other | 61

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Device Related Adverse Events.
Description: Data will be collected at the initial post-operative visit. This is a single visit study.
Time Frame: Post-op visit, after an average of 30 days
Measure: Number (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | CorMatrix ECM
Number analyzed (Participants) | 1,420
Proportion of subjects | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Data was collected through the subjects' first follow-up visit, which ranged from 0 to 229 days post-operatively.
Arm/Group | CorMatrix ECM
All-Cause Mortality (participants affected / at risk) | 8/1420
Serious Adverse Events (participants affected / at risk) | 0/1420
Other Adverse Events (participants affected / at risk) | 0/1420

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol (2014-07-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT02073331/Prot_000.pdf